CLINICAL TRIAL: NCT05210803
Title: A Long-term Follow-Up Study to Evaluate the Safety and Efficacy of Suprachoroidal Administration of RGX-314 for Participants With Neovascular Age-Related Macular Degeneration
Brief Title: Long-Term Follow-Up Study of RGX-314 Administered in the Suprachoroidal Space for Participants With nAMD
Status: Enrolling by invitation | Type: Observational
Sponsor: AbbVie (Industry)
Responsible Party: Sponsor
Other Study IDs: RGX-314-5102
Record Dates: First submitted 2022-01-14; First posted 2022-01-27 (Actual); Last update posted 2025-06-18 (Actual); Status verified 2025-06

CONDITIONS: Neovascular Age-Related Macular Degeneration (nAMD); Gene Therapy; AMD; Wet AMD; wAMD; nAMD

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Roll over: No intervention All subjects that previously received RGX-314 in a parent study
  Interventions: Other: No intervention.

INTERVENTIONS:
Other: No intervention. — All subjects that previously received RGX-314 in a parent study

SUMMARY:
This is a prospective, observational study designed to evaluate the long-term safety and efficacy of RGX-314. Eligible participants are those who were previously enrolled in a clinical study of nAMD in which they received suprachoroidal space (SCS) administration of RGX-314. Enrollment of each participant in the current study should occur after the participant has completed either the end of study or early discontinuation visit in the previous (parent) clinical study. Participants will be followed for up to 5 years after RGX-314 administration (inclusive of the parent study). As such, the total study duration for each participant may vary depending on when they enroll in the current study following RGX-314 administration in the parent study.

ELIGIBILITY:
Inclusion Criteria:

1. Must provide written, signed informed consent for this study.
2. Must have been enrolled in a previous clinical study of RGX-314 in the treatment of nAMD and must have received an SCS injection of RGX-314 in that study.
3. Must be willing and able to comply with all study procedures.

Exclusion Criteria:

1. None

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The sample sizes were determined by the parent studies and all participants who received an SCS administration of RGX-314 will be invited to participate in the long-term follow-up study. All Enrolled Population: Includes all participants who are enrolled in the long-term follow-up study.
Sampling Method: Probability Sample
Enrollment: 115 (Estimated)
Dates: Start 2021-12-20 (Actual); Primary Completion 2028-03 (Estimated); Study Completion 2028-03 (Estimated)

PRIMARY OUTCOMES:
To evaluate the long-term safety of RGX-314 | 5 years inclusive of parent study
  Incidences of ocular Adverse Events and Serious Adverse Events, and all Adverse Events of Special Interest

SECONDARY OUTCOMES:
• To evaluate the persistence of effect of RGX-314 on best corrected visual acuity (BCVA) | 5 years inclusive of parent study
  • Mean change from baseline (ie, prior to RGX-314 administration in the parent study) in BCVA
• To evaluate the persistence of effect of RGX-314 on central retinal thickness (CRT), as measured by spectral domain-optical coherence tomography (SD-OCT) | 5 years inclusive of parent study
  • Mean change from baseline (ie, prior to RGX-314 administration in the parent study) in CRT as measured by SD-OCT
• To assess the need for supplemental anti-vascular endothelial growth factor (anti-VEGF) therapy | 5 years inclusive of parent study
  • Mean number of supplemental anti-VEGF injections based on chart review
• To assess the need of clinic visits for management of nAMD | 5 years inclusive of parent study
  • Mean number of retina specialist visits attended for nAMD based on chart review

CONTACTS AND LOCATIONS:
Locations (16):
- United States (16):
  - Retinal Research Institute, LLC, Phoenix, Arizona
  - California Retina Consultants, Bakersfield, California
  - Retina-Vitreous Associates Medical Group, Beverly Hills, California
  - Northern California Retina Vitreous Associates Medical Group Inc, Mountain View, California
  - Retina Consultants San Diego, Poway, California
  - California Retina Consultants, Santa Barbara, California
  - Southeast Retina Center PC, Augusta, Georgia
  - Johns Hopkins University, Baltimore, Maryland
  - Ophthalmic Consultants of Boston, Boston, Massachusetts
  - Vitreoretinal Surgery PLLC, Edina, Minnesota
  - Sierra eye Associates, Reno, Nevada
  - Vision Research Center Eye Associates of New Mexico, Albuquerque, New Mexico
  - Retinovitreous Associates, LTD, Philadelphia, Pennsylvania
  - Charles Retina Institute, P.C, Germantown, Tennessee
  - Tennessee Retina, PC, Nashville, Tennessee
  - Retina Consultants of Texas, The Woodlands, Texas